CLINICAL TRIAL: NCT03706001
Title: Efficacy of Psychotherapy for Improving Quality of Life in Patients With Hypertrophic Cardiomyopathy and Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20182033-1
Record Dates: First submitted 2018-09-29; First posted 2018-10-15 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-09

CONDITIONS: Hypertrophic Cardiomyopathy; Depression; Anxiety; Psychotherapy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Depression; Anxiety Disorders | interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): Participants will receive psychotherapy for once a week.
  Interventions: Other: Psychotherapy
- Control Arm (No Intervention): Participants will not receive any treatment for depression.

INTERVENTIONS:
Other: Psychotherapy — Psychotherapy has gained increasing acceptance as a major treatment option for mood disorders.
  Arms: Experimental Arm

SUMMARY:
A Study to evaluate the efficacy of psychotherapy for easing the cardiac symptoms and improving and quality of life in patients with hypertrophic cardiomyopathy accompanied with depression

DETAILED DESCRIPTION:
This study will use a 8 week parallel group design. 100 patients diagnosed as hypertrophic cardiomyopathy accompanied with depression will be into experimental group and control group. The experimental group received 8 times of psychological treatments for once each week; the control group did not receive any antidepressant treatment. Follow-up assessments will be performed at baseline, week 4 and 8.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as hypertrophic cardiomyopathy;
* Diagnosed as depression;

Exclusion Criteria:

* Patients with left ventricular ejection fraction (EF) ≦ 30%;
* Renal dysfunction with serum creatinine ≧451umol/l;
* Severe heart failure and New York Heart Association (NYHA) Heart Failure Grade III;
* Combine with any type of malignant tumor;
* Combine with other serious mental illnesses such as bipolar disorder, schizophrenia, schizophrenia-like illness, severe dementia, etc.;
* Have received medication of antidepressant or psychotherapy;
* Patients with major depression; Patients with a serious risk of suicide or have had suicide attempts;
* Pregnant women and lactating women, or women who are planning to become pregnant or breastfeeding during the study period;
* Other circumstances in which the researcher judges that it is not suitable as a research object.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-10-20 (Estimated); Primary Completion 2019-09-20 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in The Quality of Life, Enjoyment and Satisfaction Questionnaire (Q-LES-Q) score between groups over time | Baseline, week 2, 4, 8
  The Quality of Life, Enjoyment and Satisfaction Questionnaire (Q-LES-Q) tests the quality of life and gives emphasis to the subjective perspective of patients on physical, psychological and social domains.

SECONDARY OUTCOMES:
Changes in The Hamilton Depression Rating Scale17 (HAM-D17) score | Baseline, week 2, 4, 8
  Hamilton Depression Rating Scale17 is a test measuring the severity of depressive symptoms in individuals. It is often used as an outcome measure of depression in research. In the 17-item version, nine of the items are scored on a five-point scale, ranging from 0 to 4. The remaining eight items are scored on a three-point scale. For the 17-item version, scores can range from 0 to 54. Scores from 0 to 6 indicate no depression, scores between 7 and 17 indicate mild depression, scores between 18 and 24 indicate moderate depression, and scores over 24 indicate severe depression.
Changes in The Hamilton Rating Scale for Anxiety (HAM-A) | Baseline, week 2, 4, 8
  The HAM-A consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Scores range from 0 to 56 where 14-17 indicates mild anxiety, 18-24 indicates moderate anxiety and scores of 25 and over indicate severe anxiety.
Changes in frequency of Syncope | Baseline, week 2, 4, 8
  A risk factor of sudden death
Changes in frequency of Arrhythmia | Baseline, week 2, 4, 8
  A risk factor of sudden death
Changes in Generalized Anxiety Disorder (GAD) -7 | Baseline, week 2, 4, 8
  A scale to test the severity of anxiety
Changes in Patient Health Questionnaire (PHQ) -9 | Baseline, week 2, 4, 8
  A scale to test the severity of depression

CONTACTS AND LOCATIONS:
Overall Officials: Liwen Liu, Doctor, Study Director — Department of Ultrasonography, Xijing Hospital, The Air Force Medical University, 127# Changle Road, Xi'an, 710032, China.; Bo Wang, Master, Study Director — Department of Ultrasonography, Xijing Hospital, The Air Force Medical University, 127# Changle Road, Xi'an, 710032, China.; Huaning Wang, Doctor, Study Chair — Department of Psychiatry, Xijing Hospital, The Air Force Medical University, 127# Changle Road, Xi'an, 710032, China.; Wenjun Wu, Master, Principal Investigator — Department of Psychiatry, Xijing Hospital, The Air Force Medical University, 127# Changle Road, Xi'an, 710032, China.

IPD SHARING:
Plan to Share IPD: Undecided
The investigator have not decided whether or not to share the data.

REFERENCES:
- [Background] Dossat AM, Sanchez-Gonzalez MA, Koutnik AP, Leitner S, Ruiz EL, Griffin B, Rosenberg JT, Grant SC, Fincham FD, Pinto JR, Kabbaj M. Pathogenesis of depression- and anxiety-like behavior in an animal model of hypertrophic cardiomyopathy. FASEB J. 2017 Jun;31(6):2492-2506. doi: 10.1096/fj.201600955RR. Epub 2017 Feb 24. PMID 28235781
- [Result] Morgan JF, O'Donoghue AC, McKenna WJ, Schmidt MM. Psychiatric disorders in hypertrophic cardiomyopathy. Gen Hosp Psychiatry. 2008 Jan-Feb;30(1):49-54. doi: 10.1016/j.genhosppsych.2007.09.005. PMID 18164940
- [Result] Igoumenou A, Alevizopoulos G, Anastasakis A, Stavrakaki E, Toutouzas P, Stefanadis C. Depression in patients with hypertrophic cardiomyopathy: is there any relation with the risk factors for sudden death? Heart Asia. 2012 Jan 1;4(1):44-8. doi: 10.1136/heartasia-2012-010099. eCollection 2012. PMID 27326027